CLINICAL TRIAL: NCT07057427
Title: Comparing the Efficacy of Nab-PHP and TCbHP in Neoadjuvant Therapy for HER2-positive Early Breast Cancer, A Multicenter, Randomized, Phase III Clinical Trial
Brief Title: Efficacy of Nab-PHP Versus TCbHP in Neoadjuvant Therapy for HER2-positive Early Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Professor, Henan Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-006Lite
Record Dates: First submitted 2025-06-24; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: HER2 positive; neoadjuvant therapy; Chemotherapy de-escalation
MeSH Terms: conditions — Breast Neoplasms | interventions — Taxes; Docetaxel; Carboplatin; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nab-PHP group (Experimental): Nab-paclitaxel(on days 1 and 8 of a 21-day cycle) + trastuzumab+ patuzumab (every 3 weeks)
  Interventions: Drug: Nab paclitaxel; Drug: Trastuzumab + Pertuzumab
- TCbHP (Active Comparator): Docetaxel + carboplatin + trastuzumab + patuzumab (every 3 weeks)
  Interventions: Drug: Docetaxel and Carboplatin; Drug: Trastuzumab + Pertuzumab

INTERVENTIONS:
Drug: Nab paclitaxel — Nab-paclitaxel (on days 1 and 8 of a 21-day cycle)
  Arms: Nab-PHP group
Drug: Docetaxel and Carboplatin — Docetaxel 75 mg/m2(day 1) + Carboplatin (AUC=6) (day 1)
  Arms: TCbHP
Drug: Trastuzumab + Pertuzumab — Trastuzumab (8mg/kg first dose, 6mg/kg sequential) and pertuzumab (840mg first dose, 420mg/kg sequential) were administered intravenously every 3 weeks, or fixed-dose combination of pertuzumab and trastuzumab for subcutaneous injection (1200 mg pertuzumab plus 600 mg trastuzumab loading dose in 15 mL, followed by 600 mg pertuzumab plus 600 mg trastuzumab maintenance doses in 10 mL), both administered every 3 weeks.

SUMMARY:
The aim of this study is to evaluate the efficacy of nab-paclitaxel (on days 1 and 8 of a 21-day cycle) compared to the standard regimen of docetaxel plus carboplatin, both combined with trastuzumab and pertuzumab, as neoadjuvant therapies for HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-70 years old.

Clinical Tumor Stage: T2-T4d, or T1c with axillary lymph node positivity.

Histologically confirmed HER2-positive invasive breast cancer:

Note: HER2 positivity is defined as at least one assessment (either initial testing or central review) by the participating center's pathology department demonstrating tumor cells with immunohistochemistry (IHC) staining intensity of 3+ or confirmation by fluorescence in situ hybridization (FISH).

Clinically measurable disease: Lesion measurable by ultrasound or MRI (optional) within 1 month prior to randomization.

Adequate organ and bone marrow function within 1 month prior to chemotherapy initiation (no contraindications to chemotherapy):

1. Absolute neutrophil count (ANC) ≥ 2.0 × 10⁹/L
2. Hemoglobin ≥ 100 g/L
3. Platelet count ≥ 100 × 10⁹/L
4. Total bilirubin < 1.5 × upper limit of normal (ULN)
5. Serum creatinine < 1.5 × ULN
6. Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) < 1.5 × ULN

Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 55% assessed by echocardiography.

Women of childbearing potential: Negative serum pregnancy test within 14 days prior to randomization.

Performance status: Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Informed consent: Provision of signed written informed consent.

Exclusion Criteria:

Stage IV (metastatic) breast cancer.

Bilateral breast cancer.

Prior systemic therapy or radiotherapy for the current breast cancer diagnosis, including chemotherapy, endocrine therapy, or targeted therapy.

History of a second primary malignancy, except for adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix.

Major surgery unrelated to breast cancer within 4 weeks prior to enrollment, or incomplete recovery from prior major surgery.

Significant cardiac disease or dysfunction, including but not limited to:

1. History of congestive heart failure or systolic dysfunction (LVEF < 50%)
2. High-risk uncontrolled arrhythmias (e.g., atrial tachycardia, resting heart rate > 100 bpm, clinically significant ventricular arrhythmia [e.g., ventricular tachycardia], or higher-grade atrioventricular block [i.e., Mobitz II second-degree or third-degree heart block])
3. Angina pectoris requiring anti-anginal medication
4. Clinically significant valvular heart disease
5. Electrocardiogram (ECG) evidence of transmural myocardial infarction
6. Poorly controlled hypertension (systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 100 mmHg)

Presence of any other severe, uncontrolled medical condition that, in the investigator's judgment, constitutes a contraindication to chemotherapy.

Known history of allergy to any component of the study drugs; patients with a history of immune deficiency diseases, including HIV positivity, or patients with other acquired or congenital immune deficiency diseases, or a history of organ transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | through study completion, up to 6 months

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | 5 years after surgery
Invasive Disease-Free Survival (iDFS) | 5 years after surgery
Safety-Number of adverse events and serious adverse events. | up to 1 year
Tolerability-Dose adjustment rate and withdrawal rate of chemotherapy drugs | up to 1 year
Residual Cancer Burden (RCB) | up to 6 months
  Proportion of patients with residual cancer burden score of 0-1 after surgery
EORTC QLQ-C30 score | up to 1 year
  quality of life evaluated by EORTC QLQ-C30
EORTC QLQ-BR23 score | up to 1 year
  quality of life evaluated by EORTC QLQ-BR23

OTHER OUTCOMES:
Exploratory endpoint - Differences in pCR rates between predefined subgroups and factors influencing pCR in the study population. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided